CLINICAL TRIAL: NCT03983967
Title: Increased Dose, Repeated Injection Clinical to Evaluate the Efficacy and Safety of 'Immuncell-LC' in Patients Undergoing Liver Transplantation With Hepatocellular Carcinoma Exceeding the Milan Criteria
Brief Title: Evaluate the Efficacy and Safety of 'Immuncell-LC' in Patients Undergoing Liver Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILC-IIT-07
Record Dates: First submitted 2019-03-12; First posted 2019-06-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Liver cancer patients undergoing liver transplantation with hepatocellular carcinoma exceeding the Milan criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuncell-LC group (Experimental): Adjuvant adoptive immune therapy using a CIK cell agent(Cytokine-Induced Killer cells; Immuncell-LC) 3 times(3 treatments at a frequency of once per week) or 6 times(3 treatments at a frequency of once per week followed by 3 treatments every 2 weeks)
  Interventions: Biological: Immuncell-LC

INTERVENTIONS:
Biological: Immuncell-LC — Activated T lymphocyte

SUMMARY:
The purpose of this study is to investigate and validate the maximum tolerated dose (MTD) or maximum available dose (MFD), safety and efficacy on patients with hepatocellular carcinoma beyond Milan criteria who undergo liver transplantation.

DETAILED DESCRIPTION:
ILC-IIT-07 is open-label, phase 1/2 clinical trial to confirm safety on patients with hepatocellular carcinoma beyond Milan criteria who undergo liver transplantation. For primary outcome, maximum feasible dose (MFD) or maximum tolerated dose (MTD) will be evaluated.

For secondary outcome, Time to Recurrence(TTR), Recurrence-Free Survival(RFS), Overall Survival(OS) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are more than 20 and less than 80 years old.
* Patients whose expected life expectancy is at least 16 weeks (4 months).
* Patients who receive liver transplants exceeding the Milan Criteria.
* ECOG Performance Status (ECOG-PS) score is 0-2.
* Patients who satisfy the following conditions of the blood test and kidney, liver function test.

Absolute neutrophil count > 500x10^6L Hemoglobin ≥ 7.5 g/dL Platelet count > 20,000/㎣ Total bilirubin < 15mg/㎗

•Patients who have agreed to participate in the study voluntarily by signing on informed consent form.

Exclusion Criteria:

* Patients who have received in vitro radiation therapy, systemic chemotherapy within 4 weeks based on sign date of Informed consent form.
* Patients who undergo ABO incompatible Liver Transplantation.
* Patients who had previously administered cell therapy.
* Patients who are confirmed with Acquired Immune Deficiency Syndrome (AIDS).
* Patients who are currently receiving dialysis.
* Patients who participated in another clinical trial and received treatment in 4 weeks or have a plan for administration of another clinical trial treatment since Informed consent form sign date.
* Patients who have uncontrollable or serious disease.
* Patients who are unable to use appropriate methods of contraception during the study period.
* Patient whose tumor has not been removed or liver metastasis is confirmed.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) or maximum feasible dose (MFD) | Every visit from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  The observation of maximum tolerated dose (MTD) or maximum feasible dose (MFD) evaluation(1X10^7cell, 5X10^7cell, 10X10^7cells) of immuncell-LC on hepatocellular carcinoma patients who undergo liver transplantation

SECONDARY OUTCOMES:
Time to Recurrence | Every visit from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  Time to Recurrence is defined as the recurring time of the cancer.
Recurrence-Free Survival | Every visit from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  Recurrence-Free Survival is defined as the recurring time of the cancer or death.
Overall Survival | Every visit from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  Overall Survival is defined as the time of death from administraion of investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Suk Suh, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No